CLINICAL TRIAL: NCT00801515
Title: A Compassionate Access Protocol For Those Patients Who Have Completed A4001029
Status: No longer available | Type: Expanded Access
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A4001090
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: HIV
Keywords: Compassionate; HIV; CCR5
MeSH Terms: interventions — Maraviroc

INTERVENTIONS:
Drug: Maraviroc — 150 mg twice per day
  Other Names: Celsentri

SUMMARY:
This is a compassionate study to provide continued access to maraviroc for only those subjects completing study A4001029 who are showing clinical benefit. Assessments of safety and tolerability of maraviroc when added to OBT will be continued.

ELIGIBILITY:
Inclusion Criteria:

* Patients having completed study A4001029 in Canada and still deriving clinical benefit.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Montreal, Quebec, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001090&StudyName=A%20Compassionate%20Access%20Protocol%20For%20Those%20Patients%20Who%20Have%20Completed%20A4001029